CLINICAL TRIAL: NCT02577653
Title: Posturographic Characteristics of Eccentric, Isometric and Concentric Movements
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics reason at the data collection site
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal investigator, Carrick Institute for Graduate Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CI-IRB-20150818005
Record Dates: First submitted 2015-10-02; First posted 2015-10-16 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: balance, postural; postural equilibrium
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subjects (Other): participant undergoing posturographic evaluation
  Interventions: Other: Posturographic evaluation

INTERVENTIONS:
Other: Posturographic evaluation — Subjects will undergo CDP testing using the modified Clinical Testing of Sensory Integration in Balance (mCTSIB) protocol. Subsequently, subjects will be asked to stand first on the right leg and then on the left leg with eyes open. Finally, subjects will be asked to perform 10 repetition of the squatting movement, with the operator pacing them (telling them when to start and when to stop the movements).

SUMMARY:
Determine the posturographic characteristics of eccentric, isometric and concentric movements in healthy subjects as well as in subjects with chronic, orthopedic conditions / pain not involving the lower extremities. The squatting movement (going down from a stand up position, bending the ankle, knee and hip joints, and then returning to the stand up position, while not lifting the feet from the supporting ground surface) is a simple motion that involves all three types of movements: eccentric (the going down), isometric (holding the down position for a couple of seconds) and concentric (the coming up). It is hypothesized that non-healthy subjects will not have "smooth" movements, and posturography could be used to separate between healthy and non-healthy subjects.

DETAILED DESCRIPTION:
Subjects will undergo Computerized Dynamic Posturography (CDP) testing using the modified Clinical Testing of Sensory Integration in Balance (mCTSIB) protocol: the subjects will be required to stand on a hard or compliant surface (a 4" tall foam cushion of known mechanical properties) in a comfortable posture, feet shoulder width, with eyes open or closed, head straight and arms to the side and free to move, gazing forward, and breathing normally. Subsequently, subjects will be asked to stand first on the right leg and then on the left leg, raising the other leg (flexing the hip about 45 degrees), bending (flexing) the knee 90 degrees, keeping the arms extended and moving them laterally (abduct shoulders to 45 degrees and extend both elbows) to help maintaining balance with eyes open. Finally, subjects will be asked to perform 10 repetition of the squatting movement, with the operator pacing them (telling them when to start and when to stop the movements). The results of the mCTSIB, combined with an initial physical and neurological examination will be used to classify the subjects into the healthy and non healthy group.

ELIGIBILITY:
Inclusion Criteria:

* subjects with chronic, orthopedic conditions / pain

Exclusion Criteria:

* involving the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Stability Score | immediately after data collection
  The Stability Score (calculated as percentage ratio of the actual sway and the theoretical limit of stability) will be used to investigate if there is any difference between healthy controls and subjects affected by chronic pain not involving the lower extremities. Statistical tools such t-tests and correlation coefficients will be used for assess if there is a difference between the two groups

SECONDARY OUTCOMES:
average velocity moment [mm^2/s] | immediately after data collection
  The average velocity moment (calculated as as the product of sway velocity path length) will be used to investigate if there is any difference between healthy controls and subjects affected by chronic pain not involving the lower extremities. Statistical tools such t-tests and correlation coefficients will be used for assess if there is a difference between the two groups
sway path length [mm] | immediately after data collection
  The sway path length (the distance traveled during the test) will be used to investigate if there is any difference between healthy controls and subjects affected by chronic pain not involving the lower extremities. Statistical tools such t-tests and correlation coefficients will be used for assess if there is a difference between the two groups
frequency content [Hz] | immediately after data collection
  The frequency content (calculated using FFT) will be used to investigate if there is any difference between healthy controls and subjects affected by chronic pain not involving the lower extremities. Statistical tools such t-tests and correlation coefficients will be used for assess if there is a difference between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Optim Orthopedics - DeRenne, Savannah, Georgia, United States